CLINICAL TRIAL: NCT03512054
Title: Pilot Study Evaluating the Success (= Safe Decannulation) of a Standardized Tracheotomy Weaning Procedure in Brain-injury's Patients
Acronym: DECATRAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2017/31
Record Dates: First submitted 2018-03-23; First posted 2018-04-30 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Tracheostomy; Brain Injuries
Keywords: Tracheostomy; Decannulation; Rehabilitation; Brain injury; Neurosurgery
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental procedure (Experimental)
  Interventions: Procedure: Standardized 5-step weaning procedure

INTERVENTIONS:
Procedure: Standardized 5-step weaning procedure — Weaning process in 5 steps (0-4), by a multi-professional team (neurosurgeon, physiotherapist, nurse, caregiver…) Stability criteria are defined for each person, after validation pass the next step. Stability criteria degradation return to the previous step. Weaning process can take back after stability criteria renormalization.
  Step 0: cuff deflate. Step 1: occlusion test. Steps 0 and 1 can assess the freedom and protect capacity airway. In failure process, we can propose a nasofibroscopy.
  Step 2: Phonatory Valve. Respiratory rehabilitation/ swallowing, limiting breathing effort. The valve ought to stay 12 hours before going to the step 3.
  Step 3: Plug. Finish the Respiratory rehabilitation/ swallowing. The plug ought to stay 24hours minimum before going to the step 4.
  Step 4: Decannulation

SUMMARY:
Tracheotomy weaning and decannulation are one of the important problems in the neurosurgical care unit. Aside from medical, psychological, sociological, economical and ethics problems, tracheotomy increases the duration of the hospital stay and conditions the secondarily future medical care (better re-education after the injury).

However, according to investigators practices, that patients who were decannulated with success can go into a secondary care residence more easily.

This research will demonstrate that all patients included can be decannulated without risk of a new recannulation in the 96 hours.

DETAILED DESCRIPTION:
Brain injury patients with alertness disorders, wake-up delay and / or swallowing disorders, frequently have a tracheotomy. This tracheotomy is often a problem when it comes to find a bed in a secondary care unit, which is better adapted to the patient rehabilitation. Unfortunately, there is little room to accept this type of patient. It is therefore appropriate to do the weaning during the neurosurgery unit stay.

Bibliographical studies indicate few recommendations as to weaning outside intensive care units. In the neurosurgery units at the University Hospital of Bordeaux, during 3 years (2014-2016), investigators have practiced 29 decannulations without recannulation, over 37 brain injury patients, with a multi-professional team (neurosurgeon, physiotherapist, nurse, caregiver…) to produce a weaning process.

From where investigators hypothesis: using a multi-professional weaning process, checking the patient's stability during the different weaning steps, can lead to decide to decannulate or not without any risk.

ELIGIBILITY:
Inclusion Criteria:

* age at least 18 years old
* brain-injury disease
* tracheotomy act while in neurosurgery or reanimation stay
* no artificial ventilation
* medical cover
* free, informed and express consent by the patient or his legal representative (no later than the day after the inclusion and before all exam necessary for the research)

Exclusion Criteria:

Malnutrition (defines by the age) :

* age < 70 years old: body mass index (B.D.I.) <16 kg/m² or albuminemia <20 g/L
* age > 70 years old: body mass index (B.D.I.) <18 kg/m² or albuminemia <30 g/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Number of safe decannulation | Up to 3 month after weaning procedure start (Inclusion)
  The main objective is to determine the effectiveness of the standardized 5-step weaning procedure for selecting patients to be decannulated without failure. This is measured by the proportion of safe decannulation for all decannulated tracheotomised patients included in the study. The failure of decannulation is defined by a recannulation within 96h.

SECONDARY OUTCOMES:
Reasons of failure in weaning process | Up to 3 month after weaning procedure start (Inclusion)
Life threatening event occurrence during the weaning procedure | Up to 3 month after weaning procedure start (Inclusion)
  Life threatening event is defined by one of the following:
  * cardiorespiratory failure,
  * septic shock,
  * cardiorespiratory arrest,
  * acute respiratory failure,
  * acute neurological condition or severe electrolyte disturbances
Mortality at 6 months | 6 month after weaning procedure start (Inclusion)
Communication capacity with CRS-R (Coma Recovery Scale Revised) communication subscore | Up 6 month after weaning procedure start (Inclusion)
  Communication subscore:
  * 2 Functional Accurate
  * 1 Non-Functional: Intentional
  * 0 None
Nutrition evolution with DOSS (Dysphagia Outcome and Severity Scale) score | Up 6 month after weaning procedure start (Inclusion)
  7 points scale:
  * Level 1: Severe dysphagia: Unable to tolerate any Per Oral safely
  * Level 7: Normal in all situations

CONTACTS AND LOCATIONS:
Overall Officials: Eric FRISON, MD, Study Chair — Unité de Soutien Méthodologique à la Recherche Clinique et Epidémiologique (USMR) du CHU de Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No